CLINICAL TRIAL: NCT04144673
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Safety and Efficacy of Bio-Active Silver Hydrosol™ in Providing Immune Support
Brief Title: A Study Investigating the Safety and Efficacy of Bio-Active Silver Hydrosol™ in Providing Immune Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immunogenics Corp. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19SIHN
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Immune Support; Active lifestyle; Silver; Healthy Adults; Cold; WURSS
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental)
  Interventions: Other: Silver Hydrosol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Silver Hydrosol — Silver quantity will be 7 doses per day, with 50 mcg per dose.
  Other Names: Sovereign Silver, Bio-Active Silver Hydrosol™
  Arms: Investigational Product
Other: Placebo — Placebo water with no active ingredients
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the ability of Bio-Active Silver Hydrosol™ in providing immune support in healthy adult males and females participating in intense aerobic exercise. Sixty eligible participants are planned to be randomized into either the investigational product or treatments arms and will consume the study product for 60 days (check-in visit on day 28). Questionnaires will be completed and blood and saliva samples will be collected to measure the endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Provided voluntary, written, informed consent to participate in the study
2. Females and males between 19 and 65 years of age inclusive
3. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening Or,

   1. Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   2. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   3. Double-barrier method
   4. Intrauterine devices
   5. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   6. Vasectomy of partner at least 6 months prior to screening
4. BMI between 18.5 to 29.9 kg/m2 inclusive
5. Individuals participating in an intense aerobic sport (e.g. cycling, running, triathlon, swimming, soccer, Nordic skiing, basketball, hockey, gym etc.) for greater than or equal to 5 hours a week
6. Agrees to provide a verbal history of flu vaccination
7. Healthy as determined by laboratory results, medical history, and physical exam or as determined by the QI
8. Agrees to maintain current diet and exercise programs
9. Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Subject has a known allergy to the test material's active or inactive ingredients
3. Verbal confirmation of a diagnosed chronic inflammatory condition
4. Verbal confirmation of the diagnosis of any autoimmune disease or immune-compromised (i.e. HIV positive, use of anti-rejection medication, rheumatoid arthritis)
5. Chronic consumption of oral anti-inflammatory medications such as cyclosporine for skin conditions such as psoriasis, dermatitis, rosacea
6. Chronic consumption of anti-inflammatory medications or medications known to affect immune function on a daily basis, including medications for allergies and asthma with the exception of Ventolin, within 4 weeks of baseline visit (visit 2)
7. Verbal confirmation of chronic recurring respiratory signs and symptoms due to allergies (including seasonal allergies) or chronic bronchitis
8. Verbal confirmation of active shingles and/or herpes virus infections, within 2 months of baseline
9. Use of medical marijuana including THC-free CBD (any form of consumption)
10. Use of recreational marijuana (any form of consumption) within the past 4 weeks and is unwilling to stop use for the duration of the study
11. Use of immunomodulators (including corticosteroids) such as immunosuppressant or immune-stimulant medications within 4 weeks of baseline
12. Taking antibiotics within 2 weeks of screening
13. Use of immune support supplements unless willing to undergo washout
14. Use of multivitamins unless on a stable regimen for 3 months as assessed by QI
15. Verbal confirmation of Type I or Type II diabetes or clinically important hepatic, cardiac, pulmonary, pancreatic, neurologic, or biliary disorder
16. History or current diagnosis of renal disease with the exception of a history of kidney stones symptom-free for 1 year
17. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
18. Current or pre-existing thyroid condition. Treatment on a stable dose medication for 6 months will be reviewed on a case-by-case basis by the QI
19. History of or current blood/bleeding disorders with the exception of a history of anemia caused by a deficiency of a mineral or vitamin, and no longer present.
20. Verbal confirmation of the diagnosis of Hepatitis B/C positive
21. Chronic unusual sleep routine (examples: irregular routine with frequent late nights, studying, partying)
22. Use of Prebiotics and Probiotics unless on a stable regimen for 3 months as assessed by QI.
23. Smoking study participants must be willing to abstain from tobacco use in the morning of a clinical visit
24. High alcohol intake (average >2 standard drinks per day, or ≥15 standard drinks per week for men, or ≥8 standard drinks per week for women)
25. Alcohol or drug abuse in the past year
26. Blood donation during or within 30 days of the last study visit
27. Subjects with unstable medical conditions as assessed by the QI
28. Clinically significant abnormal laboratory results at screening as assessed by the QI
29. Participation in a clinical research trial within 30 days prior to randomization
30. Individuals who are cognitively impaired and/or who are unable to give informed consent
31. Any other condition which in the QI's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose a significant risk to the subject

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
The difference between Bio-Active Silver Hydrosol™ and placebo in the mean global severity index, as measured by area under the curve (AUC) for the WURSS-24 daily symptom scores after 60 days supplementation. | 60 days
  The Wisconsin Upper Respiratory Symptom Survey (WURSS) is a questionnaire used to evaluate the negative impact of acute URTIs. The WURSS-24 contains 24 items scored on a Likert-type severity scale. It contains the same items as the WURSS-21 along with headache, body ache, and fever to capture influenza-like illness symptoms. The items are scored on a 0 (do not have this symptom) to 7 (severe) scale.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett B, Brown RL, Mundt MP, Thomas GR, Barlow SK, Highstrom AD, Bahrainian M. Validation of a short form Wisconsin Upper Respiratory Symptom Survey (WURSS-21). Health Qual Life Outcomes. 2009 Aug 12;7:76. doi: 10.1186/1477-7525-7-76. PMID 19674476
- See also: Explains the development of the WURSS-24 from the WURSS-21 — https://www.fammed.wisc.edu/wurss/